CLINICAL TRIAL: NCT04704141
Title: Relationship of the Gut and Genitourinary Tract Microenvironment and Male Fertility
Brief Title: Relationship of the Microenvironment and Male Fertility
Status: Not yet recruiting | Type: Observational
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Samuel Ohlander, Associate Professor of Urology, University of Illinois at Chicago
Other Study IDs: 2020-1586
Record Dates: First submitted 2021-01-07; First posted 2021-01-11 (Actual); Last update posted 2023-04-20 (Actual); Status verified 2023-04

CONDITIONS: Male Infertility; Male Hypogonadism
Keywords: Infertility; Microenvironment; Microbiome; Seminal Fluid
MeSH Terms: conditions — Infertility, Male; Eunuchism; Infertility | interventions — Hormone Replacement Therapy

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood will be collected for hormone analysis using standard analysis methods. Semen and rectal swabs will be collected and microbiome will be analyzed. All samples will be destroyed after study.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Infertile men with leukocytes in semen and eugonadal: Standard fertility evaluation and treatments
- Infertile men without leukocytes in semen and eugonadal: Standard fertility evaluation and treatments
- Infertile men with hypogonadism: Standard fertility evaluation and treatments, including hormone replacement therapy such as with clomiphene citrate
  Interventions: Drug: Hormone replacement therapy

INTERVENTIONS:
Drug: Hormone replacement therapy — A hormone replacement regimen using any medication of a number of standard treatment options
  Groups: Infertile men with hypogonadism

SUMMARY:
Although much is known about the microenvironment of the gut and the vagina, very little has been published on the microenvironment of the seminal plasma. The seminal plasma is the support fluid for sperm, providing nutrients, facilitating sperm transit to the uterus, and promoting fertilization. It is a rich area of research for markers of fertility and treatment targets.

The investigators hypothesize that (1) there are significant populations of seminal microorganisms associated with seminal leukocyte counts well below the WHO's cutoff for pyospermia (1 million/mL) that were not previously detected by traditional culturing methods, and (2) there are pathologic populations of bacteria within the gut and semen microbiome which negatively impact overall fertility, by directly or indirectly impairing hormone status.

Participants will be recruited from the Male Fertility practice at the University of Illinois-Chicago (UIC). All participants will have infertility, diagnosed as an inability to conceive pregnancy after 12 months of unprotected intercourse. The normal evaluation of these participants is to obtain at least one semen analysis and bloodwork investigating their endocrine profile: total testosterone, estradiol, sex hormone binding globulin (SHBG), luteinizing hormone (LH), follicle-stimulating hormone (FSH), and albumin. Semen volume is typically >1 mL, and <0.2 mL is typically used for the semen analysis. If over 1 million/mL round cells are identified, then a Papanicolaou stain would be performed to identify leukocytes. In this study, any semen demonstrated to have round cells would undergo Papanicolaou staining. A portion of the remaining semen, which would typically be discarded, will be sent for microbiome analysis.

Secondly, as part of routine care, fertility patients may be started on medications to increase endogenous testosterone (i.e.: clomiphene citrate, anastrozole, etc). Participants started on medications will also be asked to submit a rectal swab for gut microbiome analysis. Routine care is to monitor the hormonal and testicular response with periodic endocrine blood panels and semen analyses; rectal swabs will be requested at these follow-up intervals also. The control group for both hypotheses will be men with clinical infertility with normal semen analyses and hormone profiles.

DETAILED DESCRIPTION:
Objectives:

1. Characterize the microbiota of the genitourinary tract and testicular microenvironment in infertile men with leukocytes in the semen by using 16S rRNA sequencing to analyze the microbiome of de-identified semen samples, and compare the results of semen with normal parameters to the results of semen with leukocytes.
2. Evaluate the influence of the gut microbiome on hormone replacement therapy in hypogonadal, infertile men who are being treated with hormone replacement therapy, by analyzing multiple de-identified blood samples and rectal swabs collected both before and over the course of standard hypogonadism treatment. The investigators will use 16S rRNA sequencing on the rectal swabs and hormone level analysis of the blood samples.

Identification and Enrollment: Participants who meet inclusion criteria will be identified in UIC Urology fertility clinics by attending physician co-investigators during routine chart review for standard patient care. The participant will then be approached regarding the study and discuss the following: informed consent and information within it, basic information about the human microenvironments and significance in layman's terms, and reinforce that participation in the study will have no impact on the participant's care. Consent to participate will be obtained if the participant elects to proceed. The participant will receive oral and written information about the study. The written information includes understandable information about the study with extensive information on the study and include a copy of the consent form.

These participants' medical records will be reviewed for basic data listed below, and if hypogonadal also periodically after routine blood draws (see Venipuncture below).

Participant information management: Participants' names, MRN, and DOB will be stored in a UIC REDCap database. Each participant will also be assigned a study identification number generated by a random number generator. This ID number will be used to label the respective participant's biospecimen.

Semen collection and storage: As part of standard infertility workup of men, a semen sample will be requested after the diagnosis of infertility is made. Semen will be prospectively collected by the UIC Andrology Laboratory (820 S Wood St, Room 132, Chicago, IL 60612).

Participants will be instructed on the following for sample collection (adapted from Hou et al.):

1. Present for sample provision after 3-7 days of abstinence.
2. Wash hands 2-3 times with soap and water prior to masturbation.
3. Wash penis with a focus on glans and coronal sulcus with soap and water followed by 75% alcohol, 2-3 times.
4. Avoid contact of specimen with inside side wall of sample container.
5. 0.1 mL or less of freshly collected semen will be used for standard semen analysis.
6. If semen is identified to have any number of round cells, then a leukocyte count will be determined by Papanicolaou staining.
7. The remainder of semen will be transferred into microcentrifuge tubes, with up to 1 mL each tube, and stored in a -80C freezer within 2 hours of collection. The -80C freezer is in a locked room of the UIC Andrology Laboratory accessible to authorized personnel only.[7]

Venipuncture: Participants will have their blood drawn during standard initial evaluation of infertility. This will be performed either by UIC phlebotomy services (1801 W Taylor St Room 4B, Chicago, IL 60612) or any other phlebotomy site and laboratory based on participant preference. The endocrine profile will be determined by testing total testosterone, estradiol, sex hormone binding globulin (SHBG), luteinizing hormone (LH), follicle-stimulating hormone (FSH), and albumin levels. A total of 4.9 mL venous blood is required for these tests and thus a total of 3 gold-topped vials would be drawn from a vein. Men determined to be hypogonadal (total testosterone <300 ng/dL or bioavailable testosterone <150 ng/dL) will be requested to provide a rectal swab as well (see below). As part of standard treatment of their condition, these participants will be started on medications to increase endogenous testosterone (ie: clomiphene citrate, anastrozole, human chorionic gonadotropin, etc). Additionally, as part of standard care, these participants will be requested to return for regular assessment of medication side effects and efficacy with laboratory monitoring of their endocrine profile. This is carried out in intervals of 3-4 months at the attending physician's discretion. The laboratory data of participants meeting inclusion criteria will be recorded in a de-identified REDCap database, identified by the study ID number.

Rectal swab collection: After review of laboratory results with the participant at the first follow-up appointment, if the participant is diagnosed with infertility secondary to hypogonadism with no other identifiable causes, he will be requested to provide rectal swabs for analysis of the gut microbiome. A rectal swab kit will be provided to the participant. After a bowel movement, the participant will be asked to use the swab to collect sample from the anus and return the sample in the provided sterile plastic bag. This will be stored in a secure, locked cabinet. A rectal swab will then be requested at the same time intervals as follow-up bloodwork, collected and stored in the same manner.

Microbiota profile characterization: Microbiota analysis will be performed by the Igenomix laboratory in Valencia, Spain (Ronda Narciso Monturiol, 11 B, Parque Tecnológico Paterna, 46980 - Paterna -, Valencia, Spain). Once the investigators have prospectively collected participant samples, semen and/or rectal swabs, the investigators will periodically send samples to Igenomix for processing, as logistically feasible. The investigators will send 1 sample of each type of specimen per participant as applicable (i.e. if a participant gave enough semen for 3 additional vials in our storage freezer, then 1 vial would be sent to Igenomix; if the participant is also hypogonadal then a rectal swab is sent if it is indicated and collected as described above). Each of these samples will be identified only by study ID number and will have no PHI. Only the study ID number associated with each vial and no other identifying information will be sent with the samples, ensuring that no PHI will ever be shared with Igenomix. Igenomix laboratory will perform microbiota profiling using 16S rRNA gene sequencing in each specimen. There will be no stored samples after the analysis, as all the material will be used for DNA extraction and subsequent sequencing. All acquired data will be uploaded into a separate UIC REDCap database, with each sample's dataset identified again only by study ID number.

Data analysis: Data analysis will be performed by Dr. Pagani and UIC co-investigators to analyze the data using de-identified data sets from participant chart review and those provided by the Igenomix laboratory.

Cursory analysis of microbiota data sets will determine the exact statistical analyses applicable to address our study objectives and hypotheses. The investigators will assess bacterial microbiome composition and abundance using statistics computational programs such as the R package (R Foundation for Statistical Computing, Vienna, Austria). The investigators will further characterize the bacterial communities by creating hierarchical clustering based on published methods such as described by Hou et al. (PMID: 23993888). Based on the resulting data, the investigators will choose the appropriate statistical procedure to test our 2 hypotheses.

Study completion: Participants will be followed for 12 months, allowing for 4 follow-up appointments and sample collections. At the conclusion of our study, the investigators will destroy any remaining biospecimen. All identifiable data will be purged from the REDCap database.

ELIGIBILITY:
Inclusion Criteria:

* Men diagnosed with infertility who consent to participate in the study

Exclusion Criteria:

* Prior hormone replacement therapy
* Antibiotic use in past 6 months
* Inability to consent for self, due to age or mental capacity
* Infertility attributable to identifiable causes other than hypogonadism

Min Age: 18 Years | Sex: Male
Age Groups: Adult, Older Adult
Study Population: Males referred to University of Illinois Hospital Fertility Services
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-06 (Estimated); Primary Completion 2025-06 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Characterization of the Microbiota | 12 months
  16S rRNA sequencing of bacterial DNA found in semen and rectal swab samples will be completed on all samples obtained from participants. This will characterize the microbiota profile of each sample.

CONTACTS AND LOCATIONS:
Overall Officials: Samuel Ohlander, MD, Principal Investigator — University of Illinois at Chicago
Locations (1):
- University of Illinois Hospital, Chicago, Illinois, United States

IPD SHARING:
Plan to Share IPD: No
The investigators do not plan to make patient information available to other researchers.